CLINICAL TRIAL: NCT02151526
Title: A Phase 1/2 Open Label Study Evaluating the Safety and Efficacy of Gene Therapy of the β-Hemoglobinopathies (Sickle Cell Anemia and β-Thalassemia Major) by Transplantation of Autologous CD34+ Stem Cells Transduced Ex Vivo With a Lentiviral β-A-T87Q Globin Vector (LentiGlobin BB305 Drug Product)
Brief Title: A Study Evaluating the Safety and Efficacy of LentiGlobin BB305 Drug Product in β-Thalassemia Major (Also Referred to as Transfusion-dependent β-Thalassemia [TDT]) and Sickle Cell Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genetix Biotherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGB-205; 2012-000695-42 (EudraCT Number)
Record Dates: First submitted 2014-05-14; First posted 2014-05-30 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Beta-Thalassemia Major; Sickle Cell Disease
MeSH Terms: conditions — beta-Thalassemia; Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- LentiGlobin BB305 Drug Product (Experimental): Following myeloablative conditioning with IV busulfan for 4 consecutive days (dose may be adjusted as per protocol) and subsequent daily monitoring of busulfan levels for confirmation of adequate washout, a single dose cluster of differentiation (CD) 34+ cells/kg LentiGlobin BB305 Drug Product was administered to participants by IV infusion.
  Interventions: Drug: LentiGlobin BB305 Drug Product

INTERVENTIONS:
Drug: LentiGlobin BB305 Drug Product — LentiGlobin BB305 Drug Product was administered by intravenous (IV) infusion.

SUMMARY:
This is a Phase 1/2, open label, safety, and efficacy study of the administration of LentiGlobin BB305 Drug Product to participants with either transfusion dependent beta-thalassemia (TDT) or sickle cell disease (SCD).

ELIGIBILITY:
Inclusion Criteria:

1. Be between 5 and 35 years of age, inclusive.
2. Have severe SCD or transfusion dependent beta-thalassemia major, regardless of the genotype with the diagnosis confirmed by Hb studies. Transfusion dependence is defined as requiring at least 100 mL/kg/year of packed red blood cells (pRBCs).
3. Be eligible for allogeneic hematopoietic stem cell transplant (HSCT) based on institutional medical guidelines, but without a matched related donor.
4. Be willing and able, in the Investigator's opinion, to comply with the study procedures outlined in the study protocol.
5. Have been treated and followed for at least the past 2 years in a specialized center that maintained detailed medical records, including transfusion history.

   Participants with severe SCD also must:
6. Have failed to achieve adequate clinical benefit following hydroxyurea treatment with sufficient dosage, for at least 4 months unless this treatment was not indicated or not well tolerated.
7. Have 1 or more of the following poor prognostic risk factors:

   * Recurrent vaso occlusive crises (at least 2 episodes in the preceding year or in the year prior to start of a regular transfusion program).
   * Presence of any significant cerebral abnormality on magnetic resonance imaging (MRI) (such as stenosis or occlusions).
   * Stroke without any severe cognitive disability.
   * Osteonecrosis of 2 or more joints.
   * Anti-erythrocyte alloimmunization (>2 antibodies).
   * Presence of sickle cell cardiomyopathy documented by Doppler echocardiography.
   * Acute chest syndrome (at least 2 episodes) defined by an acute event with pneumonia-like symptoms (e.g., cough, fever [>38.5°C], acute dyspnea, expectoration, chest pain, findings upon lung auscultation, tachypnea, or wheezing) and the presence of a new pulmonary infiltrate. Participants with a chronic oxygen saturation <90% (excluding periods of SCD crisis) or carbon monoxide diffusing capacity (DLco) less than 60% in the absence of an infection should not be included in the study.
8. Participants with severe SCD and cerebral vasculopathy (defined by overt stroke; abnormal transcranial Doppler [> 170 cm/sec]; or occlusion or stenosis in the polygon of Willis; or presence of Moyamoya disease) may be enrolled only with approval by the Comite de Surveillance after review of safety and efficacy data from >or= 2 SCD participants without cerebral vasculopathy treated with LentiGlobin BB305 Drug Product

Exclusion Criteria:

1. Availability of a willing 10 /10 matched human leukocyte antigen (HLA) identical sibling hematopoietic cell donor, unless recommendation for enrollment is provided by the Comite de Surveillance following a review of the case.
2. Clinically significant, active bacterial, viral, fungal, or parasitic infection.
3. Contraindication to anesthesia for bone marrow harvesting.
4. Any prior or current malignancy, myeloproliferative or immunodeficiency disorder.
5. A white blood cell (WBC) count <3×10^9/L and/or platelet count <120×10^9/L.
6. History of major organ damage including:

   * Liver disease, with transaminase levels >3× upper limit of normal.
   * This observation will not be exclusionary if a liver biopsy shows no evidence of extensive bridging fibrosis, cirrhosis, or acute hepatitis.
   * Histopathological evidence of extensive bridging fibrosis, cirrhosis, or acute hepatitis on liver biopsy.
   * Heart disease, with a left ventricular ejection fraction <25%.
   * Kidney disease with a calculated creatinine clearance <30% normal value.
   * Severe iron overload, which in the opinion of the physician is grounds for exclusion.
   * A cardiac T2* <10 ms by magnetic resonance imaging (MRI).
   * Evidence of clinically significant pulmonary hypertension requiring medical intervention.

Ages: 5 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2013-06-07 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Antoine Ribeil, MD, Study Director — bluebird bio, Inc.
Locations (1):
- Paris, France

REFERENCES:
- [Derived] Magrin E, Semeraro M, Hebert N, Joseph L, Magnani A, Chalumeau A, Gabrion A, Roudaut C, Marouene J, Lefrere F, Diana JS, Denis A, Neven B, Funck-Brentano I, Negre O, Renolleau S, Brousse V, Kiger L, Touzot F, Poirot C, Bourget P, El Nemer W, Blanche S, Treluyer JM, Asmal M, Walls C, Beuzard Y, Schmidt M, Hacein-Bey-Abina S, Asnafi V, Guichard I, Poiree M, Monpoux F, Touraine P, Brouzes C, de Montalembert M, Payen E, Six E, Ribeil JA, Miccio A, Bartolucci P, Leboulch P, Cavazzana M. Long-term outcomes of lentiviral gene therapy for the beta-hemoglobinopathies: the HGB-205 trial. Nat Med. 2022 Jan;28(1):81-88. doi: 10.1038/s41591-021-01650-w. Epub 2022 Jan 24. PMID 35075288
- [Derived] Thompson AA, Walters MC, Kwiatkowski J, Rasko JEJ, Ribeil JA, Hongeng S, Magrin E, Schiller GJ, Payen E, Semeraro M, Moshous D, Lefrere F, Puy H, Bourget P, Magnani A, Caccavelli L, Diana JS, Suarez F, Monpoux F, Brousse V, Poirot C, Brouzes C, Meritet JF, Pondarre C, Beuzard Y, Chretien S, Lefebvre T, Teachey DT, Anurathapan U, Ho PJ, von Kalle C, Kletzel M, Vichinsky E, Soni S, Veres G, Negre O, Ross RW, Davidson D, Petrusich A, Sandler L, Asmal M, Hermine O, De Montalembert M, Hacein-Bey-Abina S, Blanche S, Leboulch P, Cavazzana M. Gene Therapy in Patients with Transfusion-Dependent beta-Thalassemia. N Engl J Med. 2018 Apr 19;378(16):1479-1493. doi: 10.1056/NEJMoa1705342. PMID 29669226
- [Derived] Ribeil JA, Hacein-Bey-Abina S, Payen E, Magnani A, Semeraro M, Magrin E, Caccavelli L, Neven B, Bourget P, El Nemer W, Bartolucci P, Weber L, Puy H, Meritet JF, Grevent D, Beuzard Y, Chretien S, Lefebvre T, Ross RW, Negre O, Veres G, Sandler L, Soni S, de Montalembert M, Blanche S, Leboulch P, Cavazzana M. Gene Therapy in a Patient with Sickle Cell Disease. N Engl J Med. 2017 Mar 2;376(9):848-855. doi: 10.1056/NEJMoa1609677. PMID 28249145

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single site in France between 07 June 2013 (First participant signed informed consent) and 26 February 2019 (Last participant last visit).
Pre-assignment Details: A total of 7 participants were treated in a single arm and completed the study. Data was planned, analyzed and reported separately for 3 participants with Sickle Cell Disease (SCD) and 4 participants with transfusion-dependent β-thalassemia (TDT).
Groups:
- LentiGlobin BB305 Drug Product for SCD: Following myeloablative conditioning with a dose (dose may be adjusted as per protocol) of 3.2 milligram per kilogram per day (mg/kg/day) busulfan intravenous (IV) for 4 consecutive days and subsequent daily monitoring of busulfan levels for confirmation of adequate washout, a single dose of greater than or equal to (> or =) 2.0×10^6 cluster of differentiation (CD) 34+ cells/kg LentiGlobin BB305 Drug Product was administered to participants with SCD by IV infusion.
- LentiGlobin BB305 Drug Product for TDT: Following myeloablative conditioning with a dose (dose may be adjusted as per protocol) of 3.2 mg/kg/day busulfan Intravenous (IV) for 4 consecutive days and subsequent daily monitoring of busulfan levels for confirmation of adequate washout, a single dose of > or =3.0 × 10^6 CD34+ cells/kg LentiGlobin BB305 Drug Product (betibeglogene autotemcel) was administered to participants with TDT by IV infusion.
Period: Overall Study
Arm/Group | LentiGlobin BB305 Drug Product for SCD | LentiGlobin BB305 Drug Product for TDT
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population consisted of all participants who initiated any study procedures, beginning with mobilization (by granulocyte-colony stimulating factor [G-CSF] with or without plerixafor) or bone marrow harvest.
Groups:
- Total: Total of all reporting groups
Arm/Group | LentiGlobin BB305 Drug Product for SCD | LentiGlobin BB305 Drug Product for TDT | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 3 | 5
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Treated Participants With Successful Neutrophil and Platelet Engraftment
Description: Neutrophil engraftment was defined as the first of absolute neutrophil count (ANC) > or = 0.5 × 10^9/ liter (L) for 3 consecutive days (or 3 consecutive measurements done on separate days), after a post-transplant value less than (<) 0.5 × 10^9/L. Platelet engraftment was defined as the first of 3 consecutive platelet values > or =20 × 10^9/L for participants with TDT and values > or =50 × 10^9/L for participants with SCD obtained on different days with no platelet transfusions administered for 7 days immediately preceding and during the evaluation period. The day of engraftment is the first day of the 3 consecutive platelet measurements.
Time Frame: From time of drug product infusion through Month 24
Population: Transplant Population (TP) included all participants in the Intent to treat population who underwent LentiGlobin BB305 Drug Product infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | LentiGlobin BB305 Drug Product for SCD | LentiGlobin BB305 Drug Product for TDT
Number analyzed (Participants) | 3 | 4
Participants
  Participants with Neutrophil Engraftment | 3 | 4
  Participants with Platelet Engraftment | 3 | 4

2. Primary Outcome: Time to Successful Neutrophil and Platelet Engraftment
Description: Neutrophil engraftment was defined as the first of ANC > or = 0.5 × 10^9/ liter (L) for 3 consecutive days (or 3 consecutive measurements done on separate days), after a post-transplant value < 0.5 × 10^9/L). Platelet engraftment was defined as the first of 3 consecutive platelet values > or =20 × 10^9/L for participants with TDT and values > or =50 × 10^9/L for participants with SCD obtained on different days with no platelet transfusions administered for 7 days immediately preceding and during the evaluation period. The day of engraftment is the first day of the 3 consecutive platelet measurements.
Time Frame: From time of drug product infusion through Month 24
Population: This outcome measure was evaluated in the Transplant Population (TP).
Measure: Median (Full Range); unit: Days
Arm/Group | LentiGlobin BB305 Drug Product for SCD | LentiGlobin BB305 Drug Product for TDT
Number analyzed (Participants) | 3 | 4
Days
  Time to Neutrophil Engraftment | 32 [27 to 38] | 16.5 [14 to 29]
  Time to Platelet Engraftment | 51 [39 to 92] | 23 [20 to 26]

3. Primary Outcome: Incidence of Transplant Related Mortality
Description: This was the safety outcome measure related to mortality. Transplant related mortality was defined as any death occurring in the study post drug product infusion deemed related to the transplant by the investigator.
Time Frame: From screening through 365 days post-transplant
Population: This outcome measure was evaluated in the Transplant Population (TP).
Measure: Number; unit: Number of deaths reported
Arm/Group | LentiGlobin BB305 Drug Product for SCD | LentiGlobin BB305 Drug Product for TDT
Number analyzed (Participants) | 3 | 4
Number of deaths reported | 0 | 0

4. Primary Outcome: Number of Participants With Overall Survival (OS) Events
Description: Overall survival was defined as time from date of LentiGlobin BB305 Drug Product infusion (Day 1) to date of death. Overall survival was censored at the date of last visit if the participant was still alive. Number of participants with OS events were reported.
Time Frame: From time of drug product infusion through Month 24
Population: Intent to Treat (ITT) population consisted of all participants who initiated any study procedures, beginning with mobilization (by Granulocyte colony stimulating factor [G-CSF] with or without plerixafor), or bone marrow harvest.
Measure: Count of Participants; unit: Participants
Arm/Group | LentiGlobin BB305 Drug Product for SCD | LentiGlobin BB305 Drug Product for TDT
Number analyzed (Participants) | 3 | 4
Participants
  Censored Participants | 3 | 4
  Participants reported OS events | 0 | 0

5. Primary Outcome: Percentage of Participants With Vector-Derived Replication-Competent Lentivirus (RCL)
Description: Blood samples were analyzed for detection of RCL using RCL co-culture assay.
Time Frame: From time of drug product infusion through Month 24
Population: This outcome measure was evaluated in the ITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | LentiGlobin BB305 Drug Product for SCD | LentiGlobin BB305 Drug Product for TDT
Number analyzed (Participants) | 3 | 4
Percentage of participants | 0 | 0

6. Primary Outcome: Number of Treated Participants With Greater Than (>) 30 Percent (%) Contribution of an Individual Clone As Per Integration Site Analysis (ISA)
Description: Clonal dominance was defined as an ISA result greater than (>) 90% of the total insertion sites (IS) at any time and a vector copy number (VCN) > or =0.3, or an initial ISA result of > 30% of the total IS with a VCN > or =0.3 followed by a result > 30% and less than or equal to (< or =) 90% at first repeat and a result > 50% at second repeat.
Time Frame: From time of drug product infusion through Month 24
Population: This outcome measure was evaluated in the Transplant Population (TP).
Measure: Count of Participants; unit: Participants
Arm/Group | LentiGlobin BB305 Drug Product for SCD | LentiGlobin BB305 Drug Product for TDT
Number analyzed (Participants) | 3 | 4
Participants | 0 | 0

7. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence associated with the use of a drug in participants, whether or not considered drug related. An AE may include a change in physical signs, symptoms, and/or clinically significant laboratory change occurring in any phase of a clinical study. This definition includes inter-current illnesses or injuries, and exacerbation of pre-existing conditions. An SAE was any AE, occurring at any dose and regardless of causality, that resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, or was considered an important medical event that may jeopardize the participant and may require medical or surgical intervention to prevent an outcome listed previously. The number of participants with AEs and SAEs were evaluated.
Time Frame: From date of Informed Consent signing up to Month 24
Population: This outcome measure was evaluated in the ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | LentiGlobin BB305 Drug Product for SCD | LentiGlobin BB305 Drug Product for TDT
Number analyzed (Participants) | 3 | 4
Participants
  Number of Participants with any Adverse Event | 3 | 4
  Number of participants with any SAE | 3 | 3

8. Secondary Outcome: Percentage of Treated Participants With Transfusion-Dependent β-Thalassemia (TDT) Who Achieved Transfusion Independence (TI)
Description: TI was defined as a weighted average hemoglobin (Hb) > or =9 grams per deciliter (g/dL) without any pRBC transfusions for a continuous period of > or =12 months at any time during the study after drug product infusion, where calculation of time period of TI starts when participants achieve a Hb > or =9 g/dL with no transfusions in the preceding 60 days.
Time Frame: From time of drug product infusion through Month 24
Population: This outcome measure was evaluated only in Transplant Population (TP) with TDT.
Measure: Number; unit: Percentage of participants
Arm/Group | LentiGlobin BB305 Drug Product for TDT
Number analyzed (Participants) | 4
Percentage of participants | 75

9. Secondary Outcome: Weighted Average Hemoglobin (Hb) During Period of Transfusion Independence (TI) in Participants With Transfusion-Dependent β-Thalassemia (TDT)
Description: as for outcome 8
Time Frame: From time of drug product infusion through Month 24
Population: This outcome measure was evaluated only in Transplant Population (TP) with TDT. The number of participants analyzed signifies participants who were evaluable for this specific outcome measure.
Measure: Median (Full Range); unit: grams per deciliter (g/dL)
Arm/Group | LentiGlobin BB305 Drug Product for TDT
Number analyzed (Participants) | 3
grams per deciliter (g/dL) | 11.3 [10.6 to 13.1]

10. Secondary Outcome: Duration of Transfusion Independence (TI) in Participants With Transfusion-Dependent β-Thalassemia (TDT)
Description: TI was defined as a weighted average Hb > or =9 grams per deciliter (g/dL) without any pRBC transfusions for a continuous period of > or =12 months at any time during the study after drug product infusion, where calculation of time period of TI starts when participants achieve a Hb > or =9 g/dL with no transfusions in the preceding 60 days. To meet the initial TI criteria, the weighted Hb must be > or =9 g/dL at the end of the 12-month period, to remain in the TI state beyond the 12-month period, the treated participant needs to maintain a weighted Hb of > or =9 g/dL from that point forward, without receiving a pRBC transfusion. This outcome measure reports the duration of TI and was evaluated in the TDT Transplant Population (TP) that reached TI.
Time Frame: From time of drug product infusion through Month 24
Population: as for outcome 9
Measure: Median (Full Range); unit: Month
Groups:
- LentiGlobin BB305 Drug Product for TDT: Following myeloablative conditioning with a dose (dose may be adjusted as per protocol) of 3.2 mg/kg/day busulfan Intravenous (IV) for 4 consecutive days and subsequent daily monitoring of busulfan levels for confirmation of adequate washout, a single dose of > or =3.0 × 10^6 CD34+ cells/kg LentiGlobin BB305 Drug Product was administered to participants with TDT by IV infusion.
Arm/Group | LentiGlobin BB305 Drug Product for TDT
Number analyzed (Participants) | 3
Month | 21.7 [21.2 to 21.8]

11. Secondary Outcome: Time From LentiGlobin BB305 Drug Product Infusion to Last Packed Red Blood Cells (pRBC) Transfusion Prior to Achieving Transfusion Independence (TI) in Participants With Transfusion-Dependent β-Thalassemia (TDT)
Description: TI was defined as a weighted average Hb > or =9 grams per deciliter (g/dL) without any pRBC transfusions for a continuous period of > or =12 months at any time during the study after drug product infusion, where calculation of time period of TI starts when participants achieve a Hb > or =9 g/dL with no transfusions in the preceding 60 days. To meet the initial TI criteria, the weighted Hb must be > or =9 g/dL at the end of the 12-month period, to remain in the TI state beyond the 12-month period, the treated participant needs to maintain a weighted Hb of > or =9 g/dL from that point forward, without receiving a pRBC transfusion. This endpoint reports the time from infusion to the last pRBC transfusion prior to achieving TI.
Time Frame: From time of drug product infusion through Month 24
Population: as for outcome 9
Measure: Median (Full Range); unit: Days
Arm/Group | LentiGlobin BB305 Drug Product for TDT
Number analyzed (Participants) | 3
Days | 11 [5 to 13]

12. Secondary Outcome: Time From LentiGlobin BB305 Drug Product Infusion to Achieving Transfusion Independence (TI) in Participants With Transfusion-Dependent β-Thalassemia (TDT)
Description: TI was defined as a weighted average Hb > or =9 grams per deciliter (g/dL) without any pRBC transfusions for a continuous period of > or =12 months at any time during the study after drug product infusion, where calculation of time period of TI starts when participants achieve a Hb > or =9 g/dL with no transfusions in the preceding 60 days. To meet the initial TI criteria, the weighted Hb must be > or =9 g/dL at the end of the 12-month period, to remain in the TI state beyond the 12-month period, the treated participant needs to maintain a weighted Hb of > or =9 g/dL from that point forward, without receiving a pRBC transfusion. This outcome measure reports the time from infusion to achievement of TI.
Time Frame: From time of drug product infusion through Month 24
Population: as for outcome 9
Measure: Median (Full Range); unit: Month
Arm/Group | LentiGlobin BB305 Drug Product for TDT
Number analyzed (Participants) | 3
Month | 14.9 [14.9 to 15.6]

13. Secondary Outcome: Weighted Average Nadir Hemoglobin (Hb) in Participants With Transfusion-Dependent β-Thalassemia (TDT)
Description: Weighted average Hb nadir was defined as an average area under the curve where the Hb closest but within 3 days prior to a transfusion was used as the Hb nadir. Hb values on the day of the transfusion were considered for nadir calculations.
Time Frame: From 6 months post-drug product infusion through Month 24
Population: This outcome measure was evaluated only in Transplant Population (TP) with TDT.
Measure: Median (Full Range); unit: grams per deciliter (g/dL)
Arm/Group | LentiGlobin BB305 Drug Product for TDT
Number analyzed (Participants) | 4
grams per deciliter (g/dL) | 11 [8.5 to 13.2]

14. Secondary Outcome: Percentage Change From Baseline in Annualized Packed Red Blood Cell (pRBC) Transfusion Volume
Description: Percent change from baseline in the average annual transfusion volume from 6 months post-drug product infusion through last visit were reported.
Time Frame: Baseline, From 6 months post-drug product infusion through Month 24
Population: This outcome measure was evaluated in the Transplant Population (TP).
Measure: Median (Full Range); unit: percent change in Annualized pRBC volume
Arm/Group | LentiGlobin BB305 Drug Product for SCD | LentiGlobin BB305 Drug Product for TDT
Number analyzed (Participants) | 3 | 4
percent change in Annualized pRBC volume | -100.0 [-100 to 90] | -100.0 [-100.0 to -100.0]

15. Secondary Outcome: Percentage Change From Baseline in Annualized Number of Packed Red Blood Cell (pRBC) Transfusions
Description: Percentage change from baseline in annualized number of pRBC transfusions from 6 months post-drug product infusion through last visit were reported.
Time Frame: Baseline, From 6 months post-drug product infusion through Month 24
Population: This outcome measure was evaluated in the Transplant Population (TP).
Measure: Median (Full Range); unit: percentage change in pRBC transfusion
Arm/Group | LentiGlobin BB305 Drug Product for SCD | LentiGlobin BB305 Drug Product for TDT
Number analyzed (Participants) | 3 | 4
percentage change in pRBC transfusion | -100.0 [-100.0 to -1.9] | -100.0 [-100.0 to -100.0]

16. Secondary Outcome: Number of Participants With Vaso-Occlusive Crisis (VOC) and/or Acute Chest Syndrome (ACS) Events Post Drug Product Infusion in Sickle Cell Disease Participants
Description: Number of VOCs, ACS, and vaso-occlusive events (VOEs; which included both VOC and ACS) through 24 months after drug product infusion.
Time Frame: From time of drug product infusion through Month 24
Population: This outcome measure was evaluated in ITT population. This outcome measure was only planned to evaluate in SCD participants. Events of VOC and ACS were from same participant.
Measure: Count of Participants; unit: Participants
Arm/Group | LentiGlobin BB305 Drug Product for SCD
Number analyzed (Participants) | 3
Participants
  Vaso-Occlusive Crisis (VOC) | 1
  Acute Chest Syndrome (ACS) | 1

17. Secondary Outcome: Therapeutic Globin Expression Measured by Hb Containing β^A -T87Q Globin (HbA^T87Q) in Peripheral Blood
Description: Therapeutic globin expression was measured by HbA^T87Q in peripheral blood and the ratio of alpha(α)- globin to all beta (β)-like-globins. The relative amount of each globin produced by a participant (including βA^A-T87Q globin) was determined in peripheral blood throughout the study.
Time Frame: From time of drug product infusion through Month 24
Population: This outcome measure was evaluated in the Transplant Population (TP).
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Arm/Group | LentiGlobin BB305 Drug Product for SCD | LentiGlobin BB305 Drug Product for TDT
Number analyzed (Participants) | 3 | 4
grams per deciliter (g/dL) | 2.947 (2.4415) | 8.287 (1.5758)

18. Secondary Outcome: Vector Copy Number (VCN) in Peripheral Blood
Description: LentiGlobin BB305 lentiviral vector (LVV) transduction efficiency was measured by VCN. The presence of vector sequences in the genomic DNA of cells is detected using quantitative polymerase chain reaction (qPCR), and results were expressed as VCN.
Time Frame: From time of drug product infusion through Month 24
Population: This outcome measure was evaluated in the Transplant Population (TP).
Measure: Mean (Standard Deviation); unit: copies per diploid genome (c/dg)
Arm/Group | LentiGlobin BB305 Drug Product for SCD | LentiGlobin BB305 Drug Product for TDT
Number analyzed (Participants) | 3 | 4
copies per diploid genome (c/dg) | 0.898 (1.1655) | 1.796 (1.3665)

ADVERSE EVENTS:
Time Frame: From date of Informed Consent signing up to Month 24
Arm/Group | LentiGlobin BB305 Drug Product for SCD | LentiGlobin BB305 Drug Product for TDT
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 3/3 | 3/4
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LentiGlobin BB305 Drug Product for SCD (N=3) | LentiGlobin BB305 Drug Product for TDT (N=4)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hepatic enzyme increased (Investigations) | 2 (2) | 0 (0)
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LentiGlobin BB305 Drug Product for SCD (N=3) | LentiGlobin BB305 Drug Product for TDT (N=4)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Xerosis (General disorders) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Puncture site pain (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 3 (8) | 4 (5)
Chills (General disorders) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Feeling cold (General disorders) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Injection site inflammation (General disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Disturbance in attention (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Premature menopause (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Catheter site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (3) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 3 (4)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 2 (2)
Staphylococcus test positive (Investigations) | 1 (1) | 0 (0)
Aspergillus test positive (Investigations) | 0 (0) | 1 (1)
Dolichocolon (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 3 (4) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 3 (15) | 4 (5)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 2 (7) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (4) | 4 (6)
Vomiting (Gastrointestinal disorders) | 3 (5) | 2 (3)
Nausea (Gastrointestinal disorders) | 3 (4) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 4 (7)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Melanoderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Folliculitis (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Genital candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Wound infection fungal (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-03-19): https://cdn.clinicaltrials.gov/large-docs/26/NCT02151526/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT02151526/SAP_001.pdf